CLINICAL TRIAL: NCT07251530
Title: Communication Enhancement Among Ventilated Patients in Intensive Care : Feasibility of Implementing "JIB-TourS cARe" High Technology Device With Eye Tracker
Brief Title: Communication Enhancement Among Ventilated Patients in Intensive Care
Acronym: CESAR
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR250036-CESAR
Record Dates: First submitted 2025-07-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Critical Care, Intensive Care
Keywords: communication; critical care; Augmentative and Alternative Communications Systems
MeSH Terms: conditions — Communication | interventions — Critical Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Communication tool for ventilated patients in intensive care — The innovative device "JIB-Tours care" is equipped with a tablet featuring eye-tracking control and software specifically dedicated to communication in an intensive care unit. The eye-tracking control allows the tablet to be used with the gaze, similar to how a computer mouse is usually used.

SUMMARY:
Intensive care is a unit that admits ventilated patients. Hospitalization is extremely challenging for these patients. Their vital prognosis is at stake, and they often have difficulty moving due to pain, edema, neuromyopathy, or the presence of monitoring cables. They are also hindered in their communication: they cannot speak because of the presence of the intubation tube between their vocal cords or the tracheostomy cannula with the inflated cuff. Every day, in each intensive care unit, about 50% of ventilated patients are conscious and face communication difficulties. They describe this difficulty as a "nightmare." This leads to challenges in care management and increases the anxiety caused by hospitalization in the intensive care unit. A large proportion of patients will develop post-intensive care syndrome. The tools currently used are not efficient. Moreover, many patients have comprehension difficulties due to the medications administered to them (sedatives) or due to the initial or secondary pathologies related to their hospitalization (confusional syndrome, ICU delirium).

Our objective is to implement an adapted and personalized communication tool for ventilated patients in intensive care.

DETAILED DESCRIPTION:
The innovative device "JIB-Tours care" is equipped with a tablet featuring eye-tracking control and software specifically dedicated to communication in an intensive care unit. The eye-tracking control allows the tablet to be used with the gaze, similar to how a computer mouse is usually used. The "JIB-Tours care" system first performs a test to assess the patient's level of understanding by analyzing eye movements. The result, provided at the end of the test, then allows the proposal of a communication interface adapted to the patient's level of understanding. Three interfaces will be available. JIB-Tours care was co-designed by intensive care healthcare professionals in collaboration with former intensive care patients and their relatives. Our objective is to evaluate the feasibility and functionality of JIB-Tours care, meaning its implementation with the patient, the completion of the understanding level test, the automated transition to the adapted communication interface, and the successful use with a message delivered by the patient in accordance with their wish.

ELIGIBILITY:
Inclusion Criteria:

* Intubated ventilated ICU patient
* Hospitalized patient with an inflated cuff tracheostomy
* conscious patient, able to open and close eyes on demand
* of-age patient
* French speaking

Exclusion Criteria:

* Patient with uncorrected visual impairment or hearing deficiency
* Known guardianship or trusteeship at the time of inclusion
* Known pregnant women at the time of inclusion and lactating patients
* opposed to the processing of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants admitted to the Intensive Care Unit of the University Hospital of Tours or Orleans or Le Mans (France)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The rate of successful uses of the "JIB-Tours care" device | Day 1
  A "successful" use is defined as (cumulative criteria, in chronological order):
  * Activation of the device by the caregiver
  * Completion of the mobility questionnaire
  * Setup of the device in front of the eligible patient
  * Successful calibration of the eye-tracking control
  * Completion of the comprehension assessment test
  * Transition to the adapted communication interface
  * Use of the communication interface by the patient by clicking on the icon requested by the caregiver

SECONDARY OUTCOMES:
Duration of device setup in front of the patient | Day 1
  This time measurement will start when the device enters the patient's room and end when the patient clicks on the requested icon. It will be timed by an independent observer.
Recording of failures according to their occurrence time | Day 1
  * Failure to start the tool
  * Failure of the mobility test
  * Failure to set up the patient
  * Failure of calibration
  * Failure to complete the comprehension test
  * Failure to transition to the adapted interface
  * Failure of communication interface operation
  * Failure during the procedure:
  * Failure due to interruption caused by patient's health status at any point in the procedure, other than a comprehension test result preventing interface proposal
Communication success rate | Day 1
  "Communication success" rate, meaning the patient successfully conveyed the intended message. The independent observer will evaluate the first message transmitted by the patient (immediately after responding to the caregiver's request to click on an icon), right after interaction with the care team. This criterion will be collected by asking the patient: "Did you succeed in conveying the information you wished to transmit?" The answer is binary: yes or no, and can be communicated by blinking, nodding, or hand squeeze. This evaluation will focus on the first message sent using the "JIB-Tours care" device.
Collection of device improvement suggestions through a feedback questionnaire from users (caregivers, patients, and relatives) | Day 28
  The independent observer will conduct individual, recorded, semi-structured interviews with patients after they have regained speech following extubation or the ability to use a phonation valve, and before discharge from intensive care. For caregivers and relatives, the semi-structured interview will be conducted immediately after device use by the independent observer. A qualitative analysis of the interviews, especially the verbatim responses, will be performed.
User satisfaction (patients, relatives, and caregivers) with the use of the "JIB-Tours care" device | Day 28
  After device use, the independent observer will present users with a scale of 4 emoticons ranging from a least smiling face to a very smiling face. The observer will ask each user to choose the emoticon that best represents their level of satisfaction with the device. The result will be recorded by the independent observer in the Case Report Form (CRF), scored from 1 (least smiling emoticon) to 4 (most smiling emoticon).

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia BODET-CONTENTIN, MD PhD, Principal Investigator — Intensive care, University Hospital, Tours
Locations (2):
- France (2):
  - Intensive care, Hospital, Le MANS, Le Mans
  - Intensive care, University Hospital, Orléans, Orléans